CLINICAL TRIAL: NCT05717855
Title: Screening of Septo-optic Dysplasia During a Fetal Examination at 16-20 Weeks of Gestation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Süleyman Salman, Associate Professor, Gaziosmanpasa Research and Education Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GaziosmanpaşaTREHu
Record Dates: First submitted 2023-01-25; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: 2D Ultrasound; Cavum Septum Pellucidum; Septooptic Dysplasia; Optic Chiasma; Willis Polygon
MeSH Terms: conditions — Septo-Optic Dysplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening septooptic dysplasia (Other): Displaying and measuring the width and length of the optic chiasm for screening septooptic dysplasia
  Interventions: Diagnostic Test: Displaying optic chiasm for screening septooptic dysplasia

INTERVENTIONS:
Diagnostic Test: Displaying optic chiasm for screening septooptic dysplasia — Displaying and measuring the width and length of the optic chiasm for screening septooptic dysplasia with ultrasound between 16-20 weeks of gestation
  Other Names: Measuring the width and length of the optic chiasm for screening septooptic dysplasia

SUMMARY:
Evaluation of prenatal optic chiasm (OC) is important for the differential diagnosis of septo-optic dysplasia (SOD), which is a congenital optic disc anomaly, and the absence of the cavum septum pellucidum (CSP). Septo-optic dysplasia is associated with a wide range of neurological abnormalities, including hypoplasia of the visual pathways, CSP agenesis, and developmental delay.

DETAILED DESCRIPTION:
Up to now, optic chiasm measurement were all done in the third trimester. in the present study, OC will be measure directly in a 2D ultrasound in coronal plane within the second trimester. In fetuses with SP agenesis, the morphology and width of the OC visual pathway may be a suitable tool to assess its development. It can also assist in the difficult task of providing prenatal counseling when faced with a diagnosis of CP agenesis. therefore In the present study, it was planned to show the optic chiasm in the screening of septooptic dysplasia by ultrasound between 16-20 weeks of gestation, and to measure the optic chiasma width and length, and to determine the mean values in the second trimester.

ELIGIBILITY:
Inclusion Criteria:

* aged greater than 18 years old
* having singleton pregnancy

Exclusion Criteria:

* being under the age of 18
* having IVF pregnancy
* having multiple pregnancy
* comorbidity during pregnancy
* smoking history
* presence of familial genetic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-03-21 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
Calculation of average width of OC according to gestational week in millimeter | 2 months
Calculation of average height of OC according to gestational week in millimeter | 2 months
Calculation of average area of OC according to gestational week millimeter square | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Turkey (Türkiye)